CLINICAL TRIAL: NCT05612100
Title: Endocrine Therapy-Induced Alopecia Natural History Evaluation Among Female Breast Cancer Survivors
Brief Title: Endocrine Therapy-Induced Alopecia in Postmenopausal and Premenopausal Female Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC220902; NCI-2022-05686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004341 (Other: Mayo Clinic Institutional Review Board); MNCCTN013 (Other: Minnesota Cancer Clinical Trials Network (MNCCTN))
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (alopecia questionnaires and surveys): Patients complete alopecia questionnaires and surveys and have medical records reviewed on study.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Other: Questionnaire Administration — Complete alopecia questionnaires
Other: Survey Administration — Complete alopecia surveys

SUMMARY:
This study evaluates endocrine therapy-induced alopecia among postmenopausal and premenopausal female patients with breast cancer. Alopecia is one of the most feared side effects of cancer-directed therapy, causing distress in women starting treatment for breast cancer. While alopecia is a well-known side effect of many chemotherapy drugs, it has also been reported by women undergoing endocrine therapy. Despite the frequent reports of alopecia related to endocrine therapy, hair loss is rarely reported as a side effect of endocrine therapy and the exact characterization of alopecia is not well understood. By having postmenopausal and premenopausal breast cancer patients describe their hair loss symptoms experienced while undergoing endocrine therapy, researchers may be able to better characterize the incidence, timing, duration, and severity of alopecia and whether the different types of endocrine therapy cause more or less trouble in this regard.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the incidence, characteristics, and severity of alopecia related to endocrine therapy in four cohorts of postmenopausal women who have had a diagnosis of breast cancer: patients undergoing endocrine therapy with tamoxifen, patients undergoing endocrine therapy with an aromatase inhibitor, patients undergoing therapy with an aromatase inhibitor in addition to a CDK4/6 inhibitor, and patients not receiving endocrine therapy. A fifth cohort has met the accrual goal and is no longer enrolling: premenopausal women receiving any type of endocrine therapy.

SECONDARY OBJECTIVE:

I. To investigate the difference in incidence, characteristics, and severity of alopecia between the aforementioned five cohorts of patients.

OUTLINE: This is an observational study.

Patients complete alopecia questionnaires and surveys and have medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Women with a diagnosis of breast cancer who are being treated with curative intent, with the one exception being women who are receiving CDK4/6 inhibitors (these patients being allowed to have more advanced disease)
* Provide informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Filling into one of the 5 groups (understanding that groups will close once they complete their accrual goals of 30 patients)
* Willingness to complete questionnaires every 3 months
* Ability to complete the first questionnaire within 2 weeks of therapy initiation (for the four arms that are receiving adjuvant hormonal therapy)

  * For patients starting tamoxifen or an aromatase inhibitor: within 2 weeks of starting tamoxifen or aromatase inhibitor
  * For patients starting a CDK 4/6 inhibitor: within 2 weeks of starting the CDK 4/6 inhibitor (patients may have started an aromatase inhibitor at any time prior to initiation of CDK 4/6 inhibitor).

Exclusion Criteria:

* Verbal baseline alopecia >= 2 on an 11 point scale (from none = 0 to severe = 10). The question to use for this item is: Please rate your hair thinning or loss on a scale from 0 to 10, with 0 being no hair loss and 10 being complete hair loss
* Planned receipt of chemotherapy or another cancer-directed therapy concurrently (e.g., everolimus, etc.; note that a CDK4/6 inhibitor is allowed within cohort 3)
* Prior use of endocrine therapy for breast cancer
* Receipt of chemotherapy over the previous 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal and premenopausal women with a diagnosis of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Estimation and characterization of patient-reported treatment-emergent alopecia within and across the cohorts | Up to study completion; up to two years
  Exact 95% confidence intervals will be created within each cohort and compared graphically using forest plots. Plots of alopecia incidence rates and severity will be plotted over time by cohort.
Overall impact on patient's quality of life | Up to study completion; up to two years
  Descriptive summaries of all the questions on the baseline and follow-up questionnaires will be tabulated to facilitate our understanding of patient-experienced alopecia and to provide a comprehensive picture of how alopecia is treated, as well as to quantify the overall impact on patient's quality of life. Standardized differences will be computed in order to give a common metric for all variables. The largest standardized difference between the pairwise cohorts will be reported.
Incidence rate of treatment-emergent alopecia | Up to study completion; up to two years
  A cumulative incidence function will be estimated in order to calculate the cumulative incidence rate (i.e. time to initial onset) of treatment-emergent alopecia, treating death and disease progression as competing risks for each cohort. Cox proportional hazards models will be used to compare differences between treatment-emergent alopecia risk between the control cohort (n=20) and the combined treatment cohorts (n = 80). The covariates included in the regression model will include age (years) and alopecia scores at baseline.
Risk of treatment-emergent alopecia | Up to study completion; up to two years
  A longitudinal analysis will be used for the binary response of whether the patient experiences treatment-emergent alopecia; this mixed model will contain an interaction between control versus treatment cohort and time, both as categorical variables, and a random intercept and slope by patient. The above covariates will also be adjusted for and piecewise splices will be used to account for any nonlinearity. The goal of the longitudinal analysis is to explore whether the risk of treatment-emergent alopecia increases with endocrine therapy exposure over time and whether this risk differs between cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cathcart-Rake, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (23):
- United States (23):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Essentia Health Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - MMCORC CentraCare Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health Moose Lake, Moose Lake, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Health Thief River Falls, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Health Worthington, Worthington, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials